CLINICAL TRIAL: NCT03340584
Title: The Effectiveness of the Nine Castle Net Format Taping After Total Knee Replacement in Early Postoperative Rehabilitation Period. A Randomized Controlled Trial
Brief Title: The Clinical Observation on Taping After Total Knee Replacement
Acronym: taping
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Song-he Jiang, Principal Investigator, Second Affiliated Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017PT1025
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Total Knee Replacement
Keywords: Total Knee Replacement; Taping; Rehabilitation; Edema; Pain
MeSH Terms: conditions — Edema; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): The intervention group will be received the Nine Castle Net Format taping and the traditional rehabilitation throughout all hospitalization period.We will exchange the new taping for Every two days.
  Interventions: Other: the Nine Castle Net Format Taping
- The control group (Other): The control group will be received the traditional rehabilitation during the hospitalization period.The traditional rehabilitation included occupational therapy and physical therapy.
  Interventions: Other: traditional rehabilitation

INTERVENTIONS:
Other: the Nine Castle Net Format Taping — The intervention group received traditional rehabilitation and Taping throughout all rehabilitation period.The taping including a Nine Castle Net Format of taping in both side of surgery knee.We will exchange the new taping for every two days， for a week.Traditional rehabilitation included occupational therapy and physical therapy, patients took part in the traditional rehabilitation training for 30 minutes each day, for a week.
  Arms: The intervention group
Other: traditional rehabilitation — traditional rehabilitation included occupational therapy and physical therapy, patients took part in the traditional rehabilitation training for 30 minutes each day, for a week.
  Arms: The control group

SUMMARY:
The investigators will conduct a single-blind, randomized controlled trial of 100 patients with total knee replacement. Patients will be randomly assigned into a control group and an intervention group.Both groups received same rehabilitation procedures after surgery,except intervention group also received taping applications throughout all rehabilitation period.Then, the patients will be reevaluated to determine changes in lower extremity function, edema, pain,knee range of motion, and muscle strength of quadriceps femoris and hamstring.

ELIGIBILITY:
Inclusion Criteria:

1. soft-tissue swelling and pain after total knee replacement
2. agree to participate the study and signing of informed consent

Exclusion Criteria:

1. severe cognitive and language barriers that can not be used to evaluate patients with pain and swelling
2. failure of important organs, such as heart, lung, liver and kidney
3. deep venous thrombosis
4. thrombophlebitis
5. varicose veins (stage II-IVaccording to Marshall) and venous insufficiency (stadium 2-3 according to Widmer)
6. participants with infection in the areas close to the knee joint, or allergy to tape
7. enrollment in another clinical trial involving physical therapy or an investigational drug

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-25 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Knee Edema at 1 week | Baseline and at 1 week
  Leg Circumference Measurements

SECONDARY OUTCOMES:
Change from Baseline Activities of Daily Living (ADL) at 1 week | Baseline and at 1 week
  The Barthel index
Change from Baseline Knee Pain at 1 week | Baseline and at 1 week
  Numeric Pain Rating Scale（NPRS）,Numeric Pain Rating Scale on a 1(no pain)to 10(worst pain imaginable)scale, 0 No pain,1 2 3 Mild pain, 4 5 6 Moderate pain,7 8 9 10 Worst possible pain
Change from Baseline Knee range of motion at 1 week | Baseline and at 1 week
  The Range of Motion Measurements
Change from Baseline muscle strength of quadriceps femoris and hamstring at 1 week | Baseline and at 1 week
  Manual Muscle Test（MMT）

CONTACTS AND LOCATIONS:
Locations (1):
- Songhe Jiang, Wenzhou, Zhejiang, China